CLINICAL TRIAL: NCT04916730
Title: Effect of Time-restricted Eating on Catecholamine-sensitivity of Adipose Tissue in Obese Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, Michael Wilkinson, Assistant Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201076
Record Dates: First submitted 2021-04-30; First posted 2021-06-07 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Key words provided by Michael Wilkinson, MD, University of California San Diego:; Catecholamine Sensitivity; Circadian Rhythm; Fasting; Obesity; Time Restricted Eating; Weight Loss
MeSH Terms: conditions — Obesity; Fasting; Intermittent Fasting; Weight Loss | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Placebo Comparator): Participants will receive standard of care nutritional behavioral counseling and will be required to log their caloric intake through the use of a smartphone app.
  Interventions: Behavioral: Standard of Care
- TRE + SOC (Experimental): Participants in this arm will receive standard of care nutritional behavioral counseling and will implement a daily, self-selected, 10-hour window within which they must consume all calories. They will also be required to log their caloric intake through the use of a smartphone app
  Interventions: Behavioral: Time Restricted Eating

INTERVENTIONS:
Behavioral: Standard of Care — Participants in this arm will receive nutritional counseling from the study dietician but will not be required to adopt a 10-hr eating window.
  Arms: Standard of Care (SOC)
Behavioral: Time Restricted Eating — Participants in this arm will adhere to a daily, consistent self-selected 10-hr eating window for the course of the study intervention period as well as receive nutritional counseling from the study dietitian.
  Arms: TRE + SOC

SUMMARY:
In a randomized controlled trial, the investigators intend to measure the health impact of time-restricted eating (TRE) in obese patients (body mass index (BMI) ≥ 30 kg/m2), who habitually eat for more than 14 hours every day. Patients will be randomly assigned to a control group of behavioral nutritional counseling (standard of care) or the intervention group of behavioral nutrition counseling with the addition of adopting a 10-hour eating window for 12 weeks (TRE).

DETAILED DESCRIPTION:
The current worldwide epidemic of obesity puts millions of people at increased risk for cardiovascular disease (CVD) and type 2 diabetes mellitus (T2DM), and while insulin resistance has been a traditional focus of treatment, resistance to catecholamines in obesity is likely a key factor hampering weight loss efforts. Catecholamines are key drivers of lipolysis in adipose tissue and bind to beta-3 adrenergic receptors (ADRB3) on the surface of adipocytes. Chronic inflammation is characteristic of obesity and suppresses the expression of adipocyte ADRB3, increasing fat storage. This leaves adipose tissue metabolically inflexible and in a state of energy preservation instead of burning fat to promote and maintain weight loss. Thus, catecholamine resistance of adipose tissue is an important target for lifestyle and therapeutic intervention. Time-restricted eating (TRE) is a therapeutic intervention that promotes weight loss and healthier metabolism by aligning dietary intake with circadian rhythms. In this RCT, individuals with obesity will be enrolled in a 14-week study of TRE and behavioral nutritional counseling vs behavioral nutritional counseling alone. In the TRE group, dietary intake will be limited to a self-selected 10-hour window. Information will be collected about adipose tissue catabolism (lipolysis) using samples collected by adipose tissue biopsy of subcutaneous abdominal adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old
2. BMI 30-50 kg/m2
3. Own a smartphone with Apple iOS or Android OS
4. Baseline eating window ≥ 14 hours/day
5. If patients are on cardiovascular medications (HMG CoA reductase inhibitors (statins), other lipid modifying drugs (including over the counter drugs such as red yeast rice and fish oil), anti-hypertensive drugs, no dose adjustments will be allowed during the study period.

Exclusion Criteria:

1. Taking insulin or anti-diabetic medications within the last 6 months.
2. Manifest diabetes, defined as fasting glucose ≥ 126 mg/dL, HbA1c ≥ 6.5%, or diagnosis of diabetes.
3. Currently taking any medication that is meant for, or has known effect on, appetite or body weight
4. Pregnant or breast-feeding women.
5. Caregiver for a dependent requiring frequent nocturnal care/sleep interruptions. Shift workers with variable (e.g. nocturnal) hours.
6. Planned international travel (time zone changes) during study period.
7. Taking therapeutic anticoagulation which might increase risk of bleeding from adipose tissue biopsy
8. History of surgical intervention for weight loss.
9. History of eating disorder
10. Currently enrolled in a weight-loss or weight-management program
11. On a special or prescribed diet for other reasons (e.g. Celiac disease)
12. Known inflammatory and/or rheumatologic disease
13. Active tobacco abuse or illicit drug use or history of treatment for alcohol abuse
14. History of bone marrow or solid organ transplant
15. History of heart failure
16. History of major adverse cardiovascular events (acute coronary syndrome (ACS), percutaneous coronary intervention, coronary artery bypass graft surgery, stroke/transient ischemic attack (TIA)).
17. History of atrial fibrillation or atrial flutter
18. History of malignancy, other than non-melanoma skin cancer, that is currently being treated, or that has not been treated with definitive therapy and considered to be in remission.
19. History of hypo- or hyperthyroidism requiring dose titration of thyroid replacement medication(s) within the past 3 months (i.e. hypothyroidism on a stable dose of thyroid replacement therapy is not an exclusion)
20. History of adrenal disease
21. History of cirrhosis
22. History of stage 4 or 5 chronic kidney disease or requiring dialysis
23. History of HIV/AIDS
24. Uncontrolled psychiatric disorder (including history of hospitalization for psychiatric illness).
25. History of obstructive sleep apnea (not on stable positive pressure therapy or other treatment for at least 3 months prior to enrollment)
26. Abnormal screening labs: renal dysfunction (eGFR < 30 ml/min/1.73 m2), anemia, hypo- or hyperthyroidism, coagulopathy, abnormal liver function (AST, ALT > 3x upper limit of normal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2026-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Wilkinson, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Altman Clinical and Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at a single academic center between November 2020 and February 2023. The first potential participant screened for study eligibility was on December 3, 2020 (enrolled (randomized) December 17, 2020) and the last participant screened for eligibility was in February 2023.
Pre-assignment Details: Out of 85 potential participants screened for study eligibility, 61 met the inclusion criteria and were subsequently randomized to treatment. One participant was excluded from analysis because of an underlying muscular dystrophy known to affect body composition.
Period: Overall Study
Arm/Group | Standard of Care (SOC) | TRE + SOC
Started | 31 | 29
Completed | 26 | 25
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | TRE + SOC | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 22 | 46
  >=65 years | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 15 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 26 | 23 | 49
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 2 | 7
  White | 18 | 20 | 38
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 29 | 60
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg^m2] | 34.7 (3.5) | 36.3 (5.9) | 35.5 (4.8)
Body Weight [Mean (Standard Deviation); unit: Kg] | 100.9 (14.7) | 101.9 (20.8) | 101.4 (17.7)

OUTCOME MEASURES:

1. Primary Outcome: Effects of TRE on Body Weight
Description: Measured as change in weight (kg).
Time Frame: Baseline to end of 12 week intervention
Population: Intent to treat population (all participants assigned to Standard of Care (SOC) or TRE + SOC).
Measure: Mean (95% Confidence Interval); unit: Kg
Arm/Group | Standard of Care (SOC) | TRE + SOC
Number analyzed (Participants) | 26 | 25
Kg | -1.68 [-2.59 to -0.77] | -4.59 [-5.51 to -3.67]
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TRE + SOC; Test type: Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Effects of TRE on Body Composition
Description: Measured as change in percent body fat.
Time Frame: Baseline to end of 12 week intervention
Measure: Mean (95% Confidence Interval); unit: percentage of body fat
Arm/Group | Standard of Care (SOC) | TRE + SOC
Number analyzed (Participants) | 25 | 25
percentage of body fat | -0.8 [-1.82 to 0.22] | -1.3 [-2.15 to -0.50]

3. Other Pre Specified Outcome: Effects of TRE on Inflammation in Obese Adipose Tissue (Exploratory Outcome)
Description: Measured as inflammatory marker mRNA.
Time Frame: Baseline to end of 12 weeks
Population: These experiments could not be conducted as planned because of budgetary constraints.
Arm/Group | Standard of Care (SOC) | TRE + SOC
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Effects of TRE on Catecholamine Sensitivity of Obese Adipose Tissue (Exploratory Outcome)
Description: Measured as release of free fatty acids (uM).
Time Frame: Baseline to end of 12 week intervention
Population: These experiments were not technically feasible with human adipose tissue
Arm/Group | Standard of Care (SOC) | TRE + SOC
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Throughout the intervention, we monitored participants for any potential adverse events.
Arm/Group | Standard of Care (SOC) | TRE + SOC
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT04916730/Prot_SAP_000.pdf